CLINICAL TRIAL: NCT04577664
Title: Total Versus Subtotal Thyroidectomy in Graves' Disease : A Randomized Controlled Trial
Brief Title: Total Versus Subtotal Thyroidectomy in Graves' Disease At AUH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Nasr, resident doctor at general surgery department, Assiut University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Thyroid surgery
Record Dates: First submitted 2020-07-28; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Thyroid Goiter
MeSH Terms: conditions — Goiter

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TT group (Active Comparator)
  Interventions: Procedure: total thyroidectomy
- ST group (Active Comparator)
  Interventions: Procedure: subtotal thyroidectomy

INTERVENTIONS:
Procedure: total thyroidectomy — a total thyroidectomy (TT) in which the entire gland is removed
  Arms: TT group
Procedure: subtotal thyroidectomy — subtotal thyroidectomy (STT) , in which most of the gland is removed leaving a small unilateral or bilateral remnant in situ about 4-5 grams.
  Arms: ST group

SUMMARY:
The main aim of work is to compare between subtotal and total thyroidectomy intra and postoperatively to identify which technique is better for patient of graves disease

DETAILED DESCRIPTION:
Graves' disease is an autoimmune disease that affects the thyroid gland[1] and it's the most common cause of hyperthyroidism. [2] Treatment of Graves' disease includes antithyroid drugs ; radioiodine ; and thyroidectomy . patients with Graves' hyperthyroidism can be treated with any of these treatment options. There is a wide geographic variation in the choice of therapy.[3] Medical treatment with antithyroid drugs is often accepted as first-choice modality in Europe, followed by radioiodine in case of recurrence. Although surgery offers the advantage of quick control and low morbidity in experienced hands, it is infrequently recommended as initial treatment. Therapy with radioiodine is the most common treatment in the United States, while antithyroid drugs and/or thyroidectomy are used more often in Europe, Japan, and most of the rest of the world.recent literature shows that the relapse rate was the highest among patients who received antithyroid drugs (40%) as compared to those who received radioiodine (21%) or Surgery (5). [4] Two different surgical techniques are used for the treatment of Graves' hyperthyroidism: a total thyroidectomy (TT) in which the entire gland is removed and a subtotal thyroidectomy (STT) , in which most of the gland is removed leaving a small unilateral or bilateral remnant in situ about 4-5 grams. Although thyroidectomy has been broadly considered as a viable alternative theapy for patients with Graves' disease , the resection extent and remnant size of thyroid gland remains controversial.[6] Although total thyroidectomy has a lower recurrence rate it has raised a concern that a more radical operation would increase the complications.[7] we intend to perform this analysis based on the published literatures of randomized controlled trials to evaluate the specific risks of thyroid surgery including recurrent hyperthyroididm , post-operative bleeding , recurrent laryngeal nerve injury , hypoparathyroidism and opthalmopathy progression.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed clinically, biochemically and immunologically with Graves' disease who will undergo thyroidectomy at general surgery department in AUH.

Exclusion Criteria:

* 1- previous thyroid or parathyroid surgery.

  * 2- recurrent hyperthyroidism after radioiodine therapy.
  * 3- preoperative recurrent laryngeal nerve palsy.
  * 4- patients unfit for operation.
  * 5- inability to comply with the follow-up protocol.
  * 6- suspicious thyroid nodules.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
comparison between total thyroidectomy vs subtotal thyroidectomy in graves' disease | baseline
  Prevlance of recurrent hyperthyroidism

SECONDARY OUTCOMES:
comparison between total thyroidectomy vs subtotal thyroidectomy in graves' disease | baseline
  Postoperative hypocalcemia and hypoparathyroidism.

REFERENCES:
- [Background] Sugino K, Nagahama M, Kitagawa W, Ohkuwa K, Uruno T, Matsuzu K, Suzuki A, Tomoda C, Y Hames K, Akaishi J, Masaki C, Ogimi Y, Yabuta T, Ito K. Change of surgical strategy for Graves' disease from subtotal thyroidectomy to total thyroidectomy: a single institutional experience. Endocr J. 2019 Feb 28;66(2):181-186. doi: 10.1507/endocrj.EJ18-0324. Epub 2018 Dec 19. PMID 30568070
- [Background] Maurer E, Maschuw K, Reuss A, Zieren HU, Zielke A, Goretzki P, Simon D, Dotzenrath C, Steinmuller T, Jahne J, Kemen M, Coerper S, Leister I, Nies C, Hartel M, Turler A, Holzer K, Agha A, Knoop M, Musholt T, Aminossadati B, Bartsch DK. Total Versus Near-total Thyroidectomy in Graves Disease: Results of the Randomized Controlled Multicenter TONIG-trial. Ann Surg. 2019 Nov;270(5):755-761. doi: 10.1097/SLA.0000000000003528. PMID 31634179
- See also: graves disease — https://www.niddk.nih.gov/health-information/endocrine-diseases/graves-disease?dkrd=hispt0296